CLINICAL TRIAL: NCT03871309
Title: Tigertriever Distal Vessels Registry
Status: Terminated | Type: Observational
Why Stopped: PI and sponsor decision
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 005-035-006-ANTR-0607
Record Dates: First submitted 2019-02-21; First posted 2019-03-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tigertriever: Male or female patients (age ≥18) who present with an acute ischemic stroke due to a M2 or distal (medium to small) vessel occlusion confirmed by vessel imaging and treated with the Tigertriever 17 or 13 revascularization devices.
  Interventions: Device: Tigertriever

INTERVENTIONS:
Device: Tigertriever — Mechanical Thrombectomy

SUMMARY:
A registry study to collect data on the Tigertriever device at restoring blood flow by removing clots in M2 or distal vessels in patients experiencing acute ischemic stroke, during commercial use.

DETAILED DESCRIPTION:
Tigertriever is a CE marked mechanical revascularization device indicated to restore blood flow by removing thrombus from a large intracranial vessel in patients experiencing ischemic stroke within 8 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with acute ischemic stroke, who can be treated within 6 hours of symptoms onset, who are either refractory to or ineligible for IV t-PA treatment and intend to be treated with thrombectomy.
* Patients ≥18
* NIHSS Score of ≥2
* Angiographically confirmed occlusion in a M2 or distal (medium to small) branch that is accessible to the Tigertriever device (17 or 13) as determined by the vessel diameter (≥1mm).
* Anticipated life expectancy of at least 6 months from presentation
* Signed informed consent form by the patient or a legally acceptable representative.

Exclusion Criteria:

* Extended infarct - ischemic changes >1/3 MCA territory / 100 ml tissue or ASPECT score <5

  * Pre- stroke mRS ≥ 2
  * Unknown time of stroke symptom onset
  * Vessel diameter < 1mm
  * Angiographically evident extreme vessel tortuosity that may preclude the device from reaching the target area.
  * Occlusion/stenosis proximal to thrombus that precludes safe retrieval
  * Medical co-morbidities including but not limited to:
  * Uncontrolled coagulopathy such as International Normalized Ratio (INR) of > 3.0 or platelets count < 40 x109/L or APTT >50 sec
  * Serious concurrent medical illness: myocardial infarction, seizures, sepsis, uncontrolled diabetes, uncontrolled hypertension, brain tumor, renal impairment (eGFR <60).
  * Baseline glucose < 2.7 or > 22.2 mmol/L
  * Imaging features of:

    * raised intracranial pressure or significant mass effect (for example, midline shift, severe sulcal effacement, transcompartmental herniation)
    * intracranial hemorrhage
    * vascular malformation or aneurysm
    * significant vascular abnormality such as carotid dissection, complete carotid occlusion or large/medium vessel vasculitis
  * Allergy/sensitivity to nickel-titanium or contrast media
  * Females who are pregnant or lactating
  * Unable to obtain informed consent from the patient or a suitable legal representative
  * Any other contraindication to thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients (age ≥18) who present with an acute ischemic stroke due to a M2 or distal (medium to small) vessel occlusion confirmed by vessel imaging and treated with the Tigertriever 17 or 13 revascularization devices.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Symptomatic Intracranial Hemorrhage (SICH) or new infarct within 24 (±12) hours post-procedure. | 24 hours post procedure
  Safety Endpoints. SICH shall be defined as Parenchymal Hematoma type 2 coupled with ≥4-point NIHSS deterioration at 24 hours.
Percentage of participants with a new occlusion. | Day 0 (end of procedure)
  Safety Endpoints.
Percentage of participants with a TICI Score ≥IIb post procedure. | Day 0 (end of procedure)
  Effectiveness Endpoints
Percentage of participants with a TICI Score ≥IIb post procedure after first pass. | Day 0 (end of procedure)
  Effectiveness Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Kyri Lobotesis, MD, Principal Investigator — Imperial College Healthcare
Locations (1):
- Imperial College Healthcare, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No